CLINICAL TRIAL: NCT02894528
Title: Evaluation of a Synthetic Bone Substitute Associated With Absorbable Collagen Membrane for Ridge Preservation After Tooth Extraction. Clinical and Tomographic Randomized Study in Humans.
Brief Title: Evaluation of a Synthetic Bone Substitute for Ridge Preservation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Sergio Luis Scombatti de Souza, Dr., University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Reprobone
Record Dates: First submitted 2016-08-24; First posted 2016-09-09 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Alveolar Process
Keywords: Alveolar ridge; guided bone regeneration; bone grafts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ridge Preservation (Test Group) (Experimental)
  Interventions: Drug: BioMend and ReproBone
- Ridge Preservation (Control Group) (Active Comparator)
  Interventions: Drug: BioMend without ReproBone

INTERVENTIONS:
Drug: BioMend and ReproBone — Post-extraction sockets was filled by synthetic bone substitute ReproBone, and after the sockets were covered by a resorbable collagen membrane BioMend, which in turn was covered by a flap.
  Arms: Ridge Preservation (Test Group)
Drug: BioMend without ReproBone — Post-extraction the socket was filled only by clot and covered by a resorbable collagen membrane BioMend, which in turn was covered by a flap.
  Arms: Ridge Preservation (Control Group)

SUMMARY:
Fifteen patients were selected, each presenting at least two jaw front teeth indicated for extraction: in the Test Group (TG), post-extraction sockets was filled by synthetic bone substitute ReproBone, and in the Control Group (CG) the socket was filled only by clot. In both groups, the sockets were covered by a resorbable collagen membrane BioMend, which in turn was covered by a flap. Computed tomography scans were acquired in the immediate postoperative period and 6 months after surgery, and the horizontal and vertical dimensional changes in bone crests were quantified.

DETAILED DESCRIPTION:
Pre-surgical procedures Before surgical procedures, all patient received oral hygiene instructions, as well as supra and subgingival root planing procedures, in order to control periodontal infections and acute inflammatory processes that could interfere with the wound healing of the sockets. Surgical procedures were performed only after the plaque index reached levels below 20%.

Surgical procedures The patients received local anesthesia (mepivacaine hydrochloride 20 mg / ml epinephrine + 0.01 mg / ml), and afther that the teeth were carefully extracted using a periotome (Hu-friedy instruments, Chicago, IL, USA). Then, vertical releasing incisions were performed in the distal faces teeths adjacent to the socket with a 15C scalpel blade, and connected by intrasulcular incisions (Figure 1b). After that, a full thickness flap was raised (Figure 1c). Granulation tissue was removed, and then clinical measurements in both selected sockets were made: Clinical Buccal Alveolar Measure (CBAM) - distance between the bottom of the socket and the buccal bone crest (Figure 1d); Clinical Palatal Alveolar Measure (CPAM) - distance between the bottom of the socket and the palatal bone crest; and Clinical Horizontal Alveolar Measure (CHAM) - distance between the buccal and palatal bone crests (Figure 1e).

Following that, in the Control Group (CG) the alveolus was filled with blood clot, while in the Test Group (TG) the alveolus was filled with a bone substitute ReproBone (Ceramisys Ltd., Sheffield,UK), (Fig. 1f). The choose between control and test sockets was randomized by a computer program (SPSS Inc., Chicago, IL, USA). The allocation of each treatment was stored in opaque envelope until immediately before the socket filling procedure.

After that, in both groups, the sockets were covered with a resorbable collagen membrane (BioMend, Zimmer Dental Inc., Carlsbad, CA, USA), which was fixed to the buccal bone plate with a titanium tack (2 mm apically to the socket bottom), which also served as a reference for tomographic measurements (Figure 1g). Then, the membrane was sutured to the lingual flap with 5-0 absorbable suture (B.Braun, Aesculap, Tuttilingen, Germany), and the flap was coronally positioned in order to cover completely the membrane (when necessary, the basis of the flap was carefully dissected to release the flap), and sutured with 4-0 silk sutures (Ethicon, Johnson & Johnson, São Paulo, Brazil), (Figure 1h). All the surgical procedures were performed by the same experimented surgeon.

Post surgical procedures All patients received systemic antibiotics (amoxycillin 500 mg, 3x day) starting 24 hours before the surgical procedure and extending for 10 days after surgery. A non-steroidal antiinflammatory drug (Nimesulide 100mg) was also prescribed, twice a day, for 5 days, as well as analgesic (750 mg paracetamol of 8/8 hours, for 3 days). A 0.12% chlorhexidine digluconate solution was prescribed as mouth rinse to be used twice a day for fifteen days. The patients were instructed to discontinue tooth brushing in the surgical area during this period. Ten days after surgery, silk sutures were removed.

A week after tooth extraction, a provisory fixed prosthesis was installed, using acrylic teeth or the crowns of the extracted teeth. Thirty days after surgery, the molding was carried out to fabricate a temporary partial denture, which was installed in all patients around 45 days after the GBR procedure; special care was taken to avoid masticatory load in the grafted area. The patients were recalled for biofilm control and reinforcement of oral hygiene instructions every 7 days in the first two months and then monthly until six months after surgery. Six months after regenerative procedure, the patients that manifested interest in oral rehabilitation with implants were referred to this service in the University.

Computerized tomographic analysis One week after surgery a Cone Bean tomography was taken (T1 - baseline) using a plastic photographic retractor (Januario et al. 2008). A single blinded calibrated (Kappa test > 80%) examiner evaluated the foolowing tomographic parameters: Tomographic Buccal Alveolar Measure (TBAM), distance between the tack and buccal alveolar crest (Figure 2); Tomographic Palatal Alveolar Measure (TPAM), distance between the tack and palatal bone crest (Figure 2); Tomographic Horizontal Apical Measure (THAM), distance between buccal and palatal bone plates, at tack level; Tomographic Horizontal Cervical Measure (THCM), distance between buccal and palatal bone plates, at crestal level (Figure 2); Tomographic Alveolar Height Measure (TAHM), distance between a line defined by the buccal and palatal bone crests and the THAM line (Figure 3).

After 6 months, a second Cone Bean tomography was taken (T2 - 6 months postoperative) as described previously. The same measures were obtained on T2 tomography in order to evaluate the dimensional changes in the period. Computerized tomography exams were acquired by a scanner model iCat Classic (Imaging Sciences International, LCC, Hatfield, PA, USA), 0.25 mm slice thickness, 0.25 mm reconstruction interval, and exposure factors of 120 KV and 36.12 mAs. Data were stored in DICOM format, and analyzed using the Ez3D Plus software.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 teeth
* Minimum of two upper front teeth with indication for extraction after clinical and radiographic examinations.

Exclusion Criteria:

* Subjects were excluded if they had systemic involvement that can interfere with periodontal treatment (e.g.: osteoporosis, diabetes, hypertension decompensated heart disease)
* Prolonged use of anti-inflammatory or steroids
* Known allergy to any biomaterial used in the study
* Smokers
* Or who were pregnant/lactating or developed this systemic condition throughout the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change the dimensions presented by the alveolar ridge after comparison of measurements at baseline and 180 days | The tomographic parameters, in millimeters, were recorded at baseline (transurgical) and 180 days after surgical procedure
  Tomographic Analysis were performed for to check the efficacy of ReproBone associated to Biomend in the preservation of the socket. The following parameters were checked: Tomographic Buccal Alveolar Measure (TBAM), distance between the tack and buccal alveolar crest; Tomographic Palatal Alveolar Measure (TPAM), distance between the tack and palatal bone crest; Tomographic Horizontal Apical Measure (THAM), distance between buccal and palatal bone plates, at tack level; Tomographic Horizontal Cervical Measure (THCM), distance between buccal and palatal bone plates, at crestal level; Tomographic Alveolar Height Measure (TAHM), distance between a line defined by the buccal and palatal bone crests and the THAM line.

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio S de Souza, Dr, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No